CLINICAL TRIAL: NCT05309655
Title: The Cardiac Outcomes With Near-Complete Estrogen Deprivation (CROWN) Study
Brief Title: Cardiac Outcomes With Near-Complete Estrogen Deprivation
Acronym: CROWN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00110774; WFBCCC 98122 (Other: Wake Forest Baptist Comprehensive Cancer Center); R01HL159393 (NIH)
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; Cardiovascular Complications
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Electrocardiography

STUDY DESIGN:
Intervention Model Description: Investigators will recruit 90 women, 67 who will be in the near-complete estrogen deprivation (NCED) group and 23 in the triple-negative breast cancer (TNBC) group. This will allow for approximately a 10% loss-to-follow-up rate and will allow investigators to have 60 participants in the NCED group and 20 in the TNBC with 2-year of data. There are 2 primary types of statistical analyses to address the study questions. The first includes testing hypotheses concerning between group (NCED vs TNBC) and within group (i.e. longitudinal changes within the NCED group) comparisons (Aims 1 and 2). The second analyses involve developing predictive equations among the NCED patients to determine if patient demographics including age, race, ethnicity, social determinants of health, clinical parameters, serum biomarkers and/or markers of inflammation are associated with cardiovascular changes over time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Near-Complete Estrogen Deprivation Therapy Participants (Experimental): Participants will receive cardiac imaging stress tests as well as study laboratory tests to monitor for changes in heart as well 30-day at the end of the study along with annual long-term follow up to 5 years from baseline imaging.
  Interventions: Drug: Adenosine Stress Cardiac Magnetic Resonance Imaging; Diagnostic Test: Electrocardiogram; Diagnostic Test: Computed Tomography Angiogram; Other: Laboratory Testing; Behavioral: Quality of Life Survey

INTERVENTIONS:
Drug: Adenosine Stress Cardiac Magnetic Resonance Imaging — Adenosine stress CMR test with contrast to include cardiovascular structural and functional measures including myocardial blood flow through quantitative perfusion mapping. Participants will have 3 stress tests as a part of this research. These tests will happen when at the beginning of the study, and then every year for 2 years.
Diagnostic Test: Electrocardiogram — A 12-lead electrocardiogram will be done when at the start of the study and at the participant's 2 year stress test to look at the electrical signals of your heart.
Diagnostic Test: Computed Tomography Angiogram — Contrasted coronary CT angiography will be performed for visual and quantitative analysis of coronary artery plaque burdens.
Other: Laboratory Testing — 10 teaspoons of blood will be withdrawn at every visit that participants receive a stress test. Participants may have up to six blood draws associated with each imaging visit.
Behavioral: Quality of Life Survey — A general health status survey with 10 questions and should take about 5-10 minutes to finish. This survey is related to research.

SUMMARY:
The purpose of this research study is to understand what effect near complete estrogen deprivation (NCED) therapy has on the heart in breast cancer patients. Investigators want to understand if NCED changes how the heart works.

DETAILED DESCRIPTION:
Primary Objective: To determine the 24-month difference in stress myocardial blood flow during adenosine stress cardiovascular magnetic resonance imaging (CMR) in premenopausal women treated with near complete estrogen deprivation for high-risk hormone receptor-positive breast cancer and in premenopausal women treated without near complete estrogen deprivation for hormone receptor-negative breast cancer.

Secondary Objectives:

* To determine the 12-month difference in stress myocardial blood flow during adenosine stress cardiovascular magnetic resonance imaging (CMR) in premenopausal women treated with near complete estrogen deprivation for high-risk hormone receptor-positive breast cancer and in premenopausal women treated without near complete estrogen deprivation for hormone receptor-negative breast cancer.
* To determine the 12-month and 24-month difference in aortic stiffness (thoracic pulse wave velocity and distensibility) with CMR in premenopausal women treated with an near complete estrogen deprivation for high-risk hormone receptor-positive breast cancer and in premenopausal women treated without near complete estrogen deprivation for hormone-receptor-negative breast cancer.
* To determine the association of stress CMR myocardial blood flow with total coronary plaque burden from coronary computed tomography angiography (at baseline and 24 month difference) and difference in variability in these measures in premenopausal women treated with near complete estrogen deprivation for high-risk hormone receptor-positive breast cancer and in premenopausal women treated without near complete estrogen deprivation for hormone receptor- negative breast cancer.
* To determine the 12-month and 24-month difference in myocardial perfusion reserve in premenopausal women treated with near complete estrogen deprivation for high-risk hormone receptor-positive breast cancer and in premenopausal women treated without near complete estrogen deprivation for hormone-receptor-negative breast cancer.
* To develop predictive models to identify women at highest risk for developing deficits in myocardial blood flow in premenopausal women treated with near complete estrogen deprivation for high-risk hormone receptor-positive breast cancer.
* To monitor disease outcomes, in particular invasive-breast cancer free survival and to assess if any changes in anti-neoplastic therapy occur on the basis cardiovascular diagnoses generally or specifically due to CROWN study results.

ELIGIBILITY:
Inclusion Criteria

* Women age ≤55 who were premenopausal at the time of breast cancer diagnosis; (Premenopausal is defined as per NCCN criteria).
* Planned breast cancer treatment with NCED (near-complete estrogen deprivation) therapy that includes aromatase inhibitor therapy (or SERD) with medically or surgically induced menopause within three (3) months of initiating NCED (HR-positive tumor) or, for the cohorts not receiving NCED therapy, within three (3) months of planned chemotherapy, surgery or radiation. Index date for three months is defined as final date of treatment with chemotherapy, surgery or radiation which ever happens last (HR-negative tumor). Treatment with a Gonadotropin Releasing Hormone (GnRH) agonist for fertility preservation during chemotherapy is allowed and is not considered part of the NCED antineoplastic therapy.
* Women with human epidermal growth factor-2 (HER2) negative and women with human epidermal growth factor-2 (HER2) positive breast cancer are eligible.
* Treatment with CDK-inhibitor, PARP inhibitor immunotherapy or biologic (non-chemotherapy) agent as part of anti-neoplastic treatment plan is allowed. These agents are not considered chemotherapy.
* Treatment with selective-estrogen receptor degrader (SERD) rather than aromatase inhibitor is allowed.
* Diagnosed with Stage I-III breast cancer.
* ECOG performance status of 0-2
* Patients with concurrent malignancies are eligible as long as therapies and disease course for these are reasonably expected to not impact cardiovascular function. (Examples of eligible malignancies include: papillary/follicular thyroid cancer, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in-situ and early stage cervical cancers, etc.).
* Patients with prior COVID-19 are eligible if they have recovered from the illness and are free of COVID-related symptoms other than allowable persistent symptoms: loss of taste and smell and/or grade 1 fatigue.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).
* The study will allow up to 30% of patients with MRI non-compatible breast expanders recognizing that baseline CMR will be outside of imaging window. Note: Registration of these participants will require study PI approval (Dr. Jordan or Dr. Thomas).

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to adenosine
* Active wheezing.
* Those with contraindications for MRI such as ferromagnetic cerebral aneurysm clips or other intracranial metal, pacemakers, defibrillators, functioning neurostimulator devices or other implanted electronic devices, or some breast expanders.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study. Because some methods of birth control are not 100% reliable, a pregnancy test is required, unless the patient has undergone either a bilateral oophorectomy, hysterectomy or both.
* Coronary revascularization in the past 6 months or known severe multi-vessel coronary artery disease previously determined to be not amendable to mechanical intervention.
* Ongoing, unrelieved symptoms thought to represent cardiac ischemia and requiring immediate cardiac catheterization
* Allergy or prior sensitivity to gadolinium or other contrasting agents or their excipients.
* Men with breast cancer.
* Known chronic renal insufficiency or chronic electrolyte abnormalities as determined by the treating physician.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Premenopausal women that are receiving or have received therapy for breast cancer.
Enrollment: 90 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Myocardial Blood Flow - 24 months | At baseline and at 24 months
  Change in myocardial blood flow will be measured by adenosine CMR imaging. Comparisons will be made using longitudinal mixed models to examine within- and between- group effects on outcomes measured. These mixed models will include fixed effects for group (NCED/TNBC), baseline assessment of the outcome of interest (i.e. MPR) to adjust for potential risk-factor profile differences between groups and the time point at which the measurements are made relative to the baseline assessment.

SECONDARY OUTCOMES:
Change in Myocardial Blood Flow - 12 months | At baseline and at 12 months
  Change in myocardial blood flow will be measured by adenosine CMR imaging. Comparisons will be made using longitudinal mixed models to examine within- and between- group effects on outcomes measured. These mixed models will include fixed effects for group (NCED/TNBC), baseline assessment of the outcome of interest (i.e. MPR) to adjust for potential risk-factor profile differences between groups and the time point at which the measurements are made relative to the baseline assessment
Change in Stiffness - Thoracic Pulse Wave Velocity | At 12 months and at 24 months
  Stiffness will be assessed by thoracic pulse wave velocity (PWV) and distensibility using CMR imaging. Comparisons will be made using longitudinal mixed models to examine within- and between- group effects on outcomes measured. These mixed models will include fixed effects for group (NCED/TNBC), baseline assessment of the outcome of interest (i.e. MPR) to adjust for potential risk-factor profile differences between groups and the time point at which the measurements are made relative to the baseline assessment
Change in Myocardial Perfusion Reserves | At 12 months and at 24 months
  Myocardial perfusion reserve will be measured with adenosine CMR imaging. Myocardial perfusion reserve is calculated as the percent change in myocardial blood flow between stress and rest perfusion imaging. Comparisons will be made using longitudinal mixed models to examine within- and between- group effects on outcomes measured. These mixed models will include fixed effects for group (NCED/TNBC), baseline assessment of the outcome of interest (i.e. MPR) to adjust for potential risk-factor profile differences between groups and the time point at which the measurements are made relative to the baseline assessment
Number of Women at High Risk for Developing Deficits in Myocardial Blood Flow | At 24 months
  The predictive models developed to identify premenopausal women treated with an aromatase inhibitor for high-risk hormone receptor-positive breast cancer at highest risk for developing deficits in myocardial blood flow will incorporate variables related to demographics, medical history, and additional clinical variables.
Overall Survival | Up to 5 years
  Disease outcomes will be monitored, including invasive-breast cancer free survival, at the annual visits throughout the study. With any change in anti-cancer therapy the specific reason for the change will be requested.
Difference in Stress CMR Myocardial Blood Flow | At baseline and at 24 months
  Total coronary plaque burden from coronary computed tomography angiography will be measured to assess the difference in heart function, including cardiac volumes and mass and blood flow in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Thomas, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Duke Cancer Center, Durham, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No